CLINICAL TRIAL: NCT05012280
Title: Malaria as a Protection Factor Against Severe COVID-19 in the Democratic Republic of Congo (Palu-COVID)
Brief Title: Malaria as a Protection Factor Against Severe COVID-19 (Known as SARS-COV-2) in the Democratic Republic of Congo (Palu-COVID)
Acronym: Palu-COVID
Status: Terminated | Type: Observational
Why Stopped: As the COVID-19 epidemic evolved, presentation of the disease changed substantially.
  Due to vaccination, increased natural immunity and new variants, there is a substantial decrease in severe cases, making it difficult to recruit new patients.
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: Palu-COVID
Record Dates: First submitted 2021-07-20; First posted 2021-08-19 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Covid19; Paludism
MeSH Terms: conditions — COVID-19; Malaria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators will explore the reasons for the apparently lower proportion of severe COVID-19 cases in many sub-Sahara African countries. Indeed, despite fragile health care systems, the burden of COVID-19 on the African continent seems substantially lower than initially feared. Many potential reasons for this discrepancy have been formulated: the different population age structure, experience of African nations with previous pandemics, warmer climate, and genetic preposition. However, another compelling hypothesis is that of trained immunity by endemic pathogens, such as plasmodia. According to this hypothesis, innate immune activation by endemic pathogens would prime a more robust initial innate immune response to SARS-CoV-2 and could therefore protect against severe COVID-19.

To explore this, the investigators propose conducting a case-control study in Kinshasa, in the Democratic Republic of the Congo (DRC). Kinshasa is an area with mixed prevalence of malaria and the area in DRC most affected by COVID-19. In this setting, the investigators will compare cases of severe COVID-19 with controls that have non-severe COVID-19 and that are matched for age, sex, and health zone. The aim is to compare pre-existing immunity against malaria, both cellular and humoral between the two groups.

ELIGIBILITY:
INCLUSION CRITERIA

To be eligible, study patients must meet the following criteria:

For cases:

* Be at least 18 years of age
* Have an RT-PCR or Antigenic Rapid Test confirmed SARS-CoV-2 infection within 72 hours prior to inclusion.
* Have given informed consent or that of their guardian/ representative to participate in the study.
* Diagnosed as a severe COVID-19 case according to the following criteria:

  * Presenting clinical signs of pneumonia: fever, cough, dyspnea or crepitations AND
  * Presenting at least one of the following signs:

Respiratory rate > 30 cycles/min OR Severe respiratory distress or SpO2 < 90% on room air

* Be admitted to a care unit for COVID-19
* Residing in the health zone for at least 6 months

For controls:

* Be at least 18 years of age
* Have a PCR or Antigenic Rapid Test-confirmed SARS-CoV-2 infection within 72 hours prior to inclusion
* Have given informed consent to participate in the study
* Diagnosed as a non-severe COVID-19 case according to the following criteria:

  * Be asymptomatic OR
  * Symptomatic, but no evidence of severe pneumonia Respiratory rate > 30 cycles/min OR Severe respiratory distress or SpO2 < 90% on room air
* Reside in the study health area for at least 6 months
* Recruited within 10 weeks following the matched cases

EXCLUSION CRITERIA

To be eligible, study patients cannot meet the following criteria for cases and controls:

* Subject has a contraindication to venipuncture, as determined by clinical judgment
* Subject is vaccinated against SARS-CoV-2
* Subject has been infected with SARS-CoV-2 in the past and now presents with reinfection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This case-control study will be conducted in the Republic of Congo in the city of Kinshasa, the epicenter of COVID-19. Kinshasa is a malaria endemic area, the distribution of malaria prevalence is lower in urban areas compared to peri-urban areas. Indeed, the city of Kinshasa is structured in four health districts and sixteen hospitals, distributed in the thirty-five Health Zones for the management of COVID-19.
  The study will consist of cases and controls:
  * Cases will be severe COVID-19 cases that will consist of patients hospitalized and recruited in COVID-19 Treatment Centers.
  * Controls will consist of asymptomatic or symptomatic cases without signs of severity. For each case, two controls will be recruited after having been matched in terms of age, gender and health zone of origin.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut National De Recherche Biomédical (INRB), Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 137 cases and 101 controls were included in the trial. Total paired matched case-controls at the end of study: 95 (95 controls and 95 cases).
  Baseline characteristics were entered for the matched case-control participants.
Groups:
- Cases: Cases are severe COVID-19 cases and comprise inpatients recruited from CTCOs.
  * Presenting clinical signs of pneumonia: fever, cough, or respiratory difficulties AND
  * Presenting at least one of the following:
    * Respiratory rate > 30 breaths/min OR
    * Severe respiratory distress (clarification: with oxygen) OR
    * SpO2 < 90% in room air (clarification: without oxygen)
  * Be admitted to a care unit for COVID-19 (clarification: hospital)
- Controls: Controls are asymptomatic or symptomatic cases without signs of severity:
  * Asymptomatic OR
  * Symptomatic, but without any signs of severe pneumonia:
    * Respiratory rate ≤ 30 breaths/min AND
    * No severe respiratory distress AND
    * SpO2 ≥ 90% in room air
  * Recruited within 10 weeks of a matched case
Period: Overall Study
Arm/Group | Cases | Controls
Started | 137 | 101
Completed | 137 | 97
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 95 | 95 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 73 | 138
  >=65 years | 30 | 22 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [40 to 66] | 54 [38 to 63] | 55 [38 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 112
  Male | 39 | 39 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 95 | 95 | 190
Civil status [Count of Participants; unit: Participants]
  Single | 18 | 22 | 40
  Married | 63 | 51 | 114
  Widow(er) | 14 | 19 | 33
  No information | 0 | 3 | 3
Level of education [Count of Participants; unit: Participants]
  Illiterate | 4 | 1 | 5
  Primary school degree | 14 | 13 | 27
  Secondary school degree | 37 | 44 | 81
  Higher education/university | 38 | 37 | 75
  No information | 2 | 0 | 2
Occupation [Count of Participants; unit: Participants]
  No job occupation | 45 | 30 | 75
  farmer | 1 | 3 | 4
  Maintenance worker | 1 | 1 | 2
  driver | 1 | 7 | 8
  Shopkeeper/Store clerk | 10 | 10 | 20
  Office worker/Public servant | 11 | 11 | 22
  teacher | 5 | 7 | 12
  gardener | 0 | 1 | 1
  worker | 0 | 2 | 2
  technician | 4 | 2 | 6
  other | 14 | 21 | 35
  no information | 3 | 0 | 3
Health Zone of Kinshasa [Count of Participants; unit: Participants]
  Bandalungwa | 2 | 2 | 4
  Barumbu | 1 | 1 | 2
  Binza-Meteo | 1 | 1 | 2
  Binza-Ozone | 4 | 4 | 8
  Gombe | 5 | 5 | 10
  Kalamu I | 1 | 1 | 2
  Kalamu II | 1 | 1 | 2
  Kasa-Vubu | 2 | 2 | 4
  Kimbanseke | 7 | 7 | 14
  Kintambo | 2 | 2 | 4
  Kisenso | 2 | 2 | 4
  Lemba | 14 | 14 | 28
  Limete | 12 | 12 | 24
  Lingwala | 1 | 1 | 2
  Makala | 1 | 1 | 2
  Masina I | 5 | 5 | 10
  Masina II | 2 | 2 | 4
  Matete | 4 | 4 | 8
  Mont-Ngafula I | 8 | 8 | 16
  Ndjili | 1 | 1 | 2
  Ngaba | 2 | 2 | 4
  Ngiri-Ngiri | 3 | 3 | 6
  Nsele | 13 | 13 | 26
  Selembao | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Malaria Antibody Level
Description: Malaria antibody level in severe and non-severe COVID-19 cases. This level will be assessed by measuring the concentration of IgG against Circum Sporozoite Protein (CSP) using the Luminex- MAGPIX, which is expressed in fluorescence intensity.
  Analysis of Conditional Maximum Likelihood Estimates.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: fluorescence intensity (log scale)
Groups:
- Cases: The cases will be severe COVID-19 cases, and will comprise hospitalized patients recruited from COVID-19 Treatment Centers.
- Controls: Controls will consist of asymptomatic or symptomatic COVID-19 cases without signs of severity.
Arm/Group | Cases | Controls
Number analyzed (Participants) | 95 | 95
fluorescence intensity (log scale) | 3.8 [2.4 to 4.7] | 3.3 [2.6 to 4.5]
Statistical Analysis 1: Comparison: Cases; Test type: Superiority; p = 0.1150, Regression, Logistic — only one primary endpoint, p value not adjusted for multiple comparisons. A priori treshold or statistical significance: p=0.05; conditional logistic regression for matched case control; Odds Ratio (OR) = 1.221, 95% CI 2-sided [0.953 to 1.564]
Statistical Analysis 2: Comparison: Cases vs Controls; Test type: Superiority; p = 0.12, Regression, Logistic; conditional logistic regression for matched case control study; Odds Ratio (OR) = 1.221, 95% CI 2-sided [0.953 to 1.564]

ADVERSE EVENTS:
Time Frame: no adverse events or deaths collected as it is not applicable (no investigational product)
Description: no adverse events or deaths collected as it is not applicable (no investigational product)
Arm/Group | Cases | Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT05012280/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT05012280/SAP_001.pdf